CLINICAL TRIAL: NCT04191629
Title: Phase 1 Clinical Study to Evaluate Safety and Tolerability of Magnetic Human Corneal Endothelial Cells in the Treatment of Corneal Edema
Brief Title: Phase 1 Study to Evaluate the Safety and Tolerability of EO1404 in the Treatment of Corneal Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valeria Sanchez-Huerta (Other)
Collaborators: Emmecell (Industry)
Responsible Party: Sponsor-Investigator, Valeria Sanchez-Huerta, Academic Director, Asociación para Evitar la Ceguera en México
Organization: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VSH01
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Corneal Edema; Fuchs Dystrophy; Fuchs' Endothelial Dystrophy; Pseudophakic Bullous Keratopathy; Corneal Endothelial Dystrophy; Corneal Transplant Failure
MeSH Terms: conditions — Corneal Edema; Fuchs' Endothelial Dystrophy; Corneal Dystrophy, Posterior Polymorphous, 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50K to 200K cells (Experimental)
  Interventions: Combination Product: EO1404
- 50K to 200K cells with endothelial brushing (Experimental)
  Interventions: Combination Product: EO1404; Procedure: Endothelial brushing or Descemet stripping
- 500K cells (Experimental)
  Interventions: Combination Product: EO1404
- 500K cells with endothelial brushing (Experimental)
  Interventions: Combination Product: EO1404; Procedure: Endothelial brushing or Descemet stripping

INTERVENTIONS:
Combination Product: EO1404
  Other Names: Magnetic Human Corneal Endothelial Cells
Procedure: Endothelial brushing or Descemet stripping
  Arms: 500K cells with endothelial brushing; 50K to 200K cells with endothelial brushing

SUMMARY:
Single center, phase 1 study to evaluate the safety and tolerability of EO1404 in subjects with corneal edema secondary to pseudophakic bullous keratopathy or Fuch's endothelial dystrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Pseudophakic with a posterior chamber intraocular lens.
3. Symptomatic corneal edema associated with endothelial dysfunction which may be secondary to Fuchs corneal dystrophy or pseudophakic bullous keratopathy.

   a Symptoms including reduced vision and/or glare, and/or pain; subject may or may not have been on topical therapies such as 5% sodium chloride drops or prednisolone acetate 1% drops.

   b ETDRS-best corrected visual acuity worse than 20/63 on Snellen. c Central corneal thickness < 2 mm by ultrasound pachymetry or OCT. d Subject must have progressed far enough in their clinical course to be considered a surgical candidate for full-thickness corneal transplantation or endothelial keratoplasty.
4. Subject must understand and sign the informed consent. If the subject's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the subject in their maternal language.
5. Subject must be medically able and willing to undergo the protocol-required procedures.

Exclusion Criteria:

All ocular criteria apply to study eye unless otherwise noted.

1. Other corneal disease, including active or prior herpetic ocular infection; active inflammation; corneal scarring from trauma, burns, or infection; or band keratopathy.
2. Visual acuity in the fellow eye is worse than 20/200.
3. Anterior chamber intraocular lens.
4. Subject requires topical, intravenous or oral acyclovir and/or related products during study duration
5. History of vitrectomy.
6. History of refractive surgery.
7. Macular disease that in the investigator and/or sponsor's opinion would limit the ability of the subject to demonstrate improvement in BCVA.
8. Prior incisional eye surgery within 3 months prior to study treatment.
9. Subject is receiving systemic steroids or other systemic immunosuppressive medications.
10. Subject is currently participating in or has participated within the last 3 months in any other clinical trial of an investigational drug by ocular or systemic administration.
11. History of uveitis or other ocular inflammatory disease.
12. History of glaucoma, or peripheral anterior synechiae on gonioscopy.
13. History of incisional glaucoma surgery (e.g., trabeculectomy, glaucoma drainage implant).
14. Female subject who is pregnant, nursing, or planning to become pregnant, or who is of childbearing potential and not using a reliable means of contraception during the study.
15. Subject is immunodeficient, or tested positive for HIV.
16. Subject is on chemotherapy.
17. History of malignancy other than basal cell carcinoma, UNLESS the malignancy was treated successfully 5 years prior to inclusion in the study.
18. History of ocular neoplasm.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-05-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Adverse Events | 12 months
  Evaluation of safety adverse events including worsening of corneal edema and increase in intraocular pressure

SECONDARY OUTCOMES:
BVCA | 12 months
  Best corrected visual acuity
Corneal thickness | 12 months
  Decrease in corneal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Sanchez-Huerta, MD, Principal Investigator — Asociacion Para Evitar la Ceguera
Locations (1):
- Asociación Para Evitar la Ceguera en México, IAP, Hospital "Dr. Luis Sánchez Bulnes", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No